CLINICAL TRIAL: NCT05814718
Title: Multicenter Randomized Controlled Clinical Study of Mitoxantrone Hydrochloride Liposome Injection Combined With Carmustine, Etoposide and Cytarabine (Modified BEAM Protocol) for T Cell Lymphoma Underwent Autologous Stem Cell Transplantation
Brief Title: Modified BEAM Regimen for T Cell Lymphoma Underwent ASCT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: First Affiliated Hospital Xi'an Jiaotong University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: XJTU1AF2022LSL-018
Record Dates: First submitted 2023-02-22; First posted 2023-04-18 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: Autologous Stem Cell Transplantation; Conditioning
MeSH Terms: interventions — Carmustine; Cytarabine; Etoposide; Melphalan

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- modified BEAM conditioning regimen (Experimental): Mitoxantrone liposome 24 mg/m2，ivgtt，d-7；BCNU 300 mg/m2，ivgtt，d-6； Ara-C 200 mg/m2 q12h，ivgtt，d-5- -2； Vp16 200 mg/m2 ，ivgtt，d-5- -2；
  Interventions: Drug: modified BEAM
- BEAM conditioning regimen (Active Comparator): BCNU 300 mg/m2，-7d； Vp16 200 mg/m2，-6～-3d； Ara-C 100mg/m2 q12h，-6～-3d； Mel 140mg/m2，-2d
  Interventions: Drug: BEAM

INTERVENTIONS:
Drug: modified BEAM — Mitoxantrone liposome 24 mg/m2，ivgtt，d-7；BCNU 300 mg/m2，ivgtt，d-6； Ara-C 200 mg/m2 q12h，ivgtt，d-5- -2； Vp16 200 mg/m2 ，ivgtt，d-5- -2；
  Other Names: Mitoxantrone liposome; Carmustine; Cytarabine; Etoposide
  Arms: modified BEAM conditioning regimen
Drug: BEAM — BCNU 300 mg/m2，-7d； Vp16 200 mg/m2，-6～-3d； Ara-C 100mg/m2 q12h，-6～-3d； Mel 140mg/m2，-2d
  Other Names: Carmustine; Cytarabine; Etoposide; Melphalan
  Arms: BEAM conditioning regimen

SUMMARY:
A multicenter randomized study on the efficacy and safety of mitoxantrone hydrochloride liposome injection combined with carmustine, etoposide, and cytarabine (modified BEAM protocol) in the pretreatment of T-cell lymphoma underwent autologous stem cell transplantation

DETAILED DESCRIPTION:
T-cell lymphoma patients with the indication of autologous stem cell transplantation will be divided into two groups，the control group will use BEAM as conditioning regimen and the experiment group will use modified BEAM regimen（included mitoxantrone liposome，then to compare the efficacy and safety of the two conditioning regimens for patients.

ELIGIBILITY:
Inclusion Criteria:

* 1) Subjects volunteered to participate in the study, signed the informed consent form, had good compliance and cooperated with follow-up 2) 18~60 years old (including upper and lower limits) 3) Patients who were pathologically diagnosed as T-cell lymphoma and planned to undergo autologous hematopoietic stem cell transplantation 4) ECOG score 0-1 5) Organ function level must meet the following requirements:

  1. Liver: aspartate aminotransferase (AST), alanine aminotransferase (ALT) ≤ 3 times the upper limit of normal (ULN), total bilirubin (TBIL) ≤ 1.5 × ULN (AST, ALT ≤ 5 is allowed in case of liver invasion × ULN）；
  2. Kidney: blood creatinine ≤ 1.5 × ULN；
  3. Coagulation function: International normalized ratio (INR) and activated partial thromboplastin time (APTT) ≤ 1.5 × ULN；
  4. Normal cardiac function: normal or abnormal ECG, no clinical significance, left ventricular ejection fraction (LVEF) shown by cardiac ultrasound is greater than 60, or myocardial zymogram CK-MB is normal, and pro BNP is less than 900 pg/ml 6) The serum pregnancy test results of female subjects with reproductive capacity must be negative before the first use of the test drug

Exclusion Criteria:

* 1.The previous anti-tumor treatment history of the subject meets one of the following conditions:

  1. Those who have previously received mitoxantrone or mitoxantrone liposomes
  2. Have received doxorubicin or other anthracyclines before, and the total cumulative dose of doxorubicin is more than 360 mg/m2 (1 mg doxorubicin equivalent to 2 mg epirubicin for other anthracyclines) 2. Hypersensitivity to any study drug or its components 3. Uncontrollable systemic diseases (such as active infection, uncontrollable hypertension, diabetes, etc.) 4. Heart function and disease meet one of the following conditions:

  <!-- -->

  1. Long QTc syndrome or QTc interval>480 ms
  2. Complete left bundle branch block, grade II or III atrioventricular block
  3. Serious and uncontrolled arrhythmia requiring drug treatment
  4. American New York Heart Association rating ≥ III
  5. Cardiac ejection fraction (LVEF) is less than 60%
  6. A history of myocardial infarction, unstable angina, severe unstable ventricular arrhythmia or any other arrhythmia requiring treatment, a history of clinically serious pericardial disease, or ECG evidence of acute ischemia or active conduction system abnormality within 6 months before recruitment.

     5. Active infection of hepatitis B and hepatitis C (hepatitis B virus surface antigen is positive and hepatitis B virus DNA exceeds 1x103 copies/mL, hepatitis C virus RNA exceeds 1x103 copies/mL) 6. Human immunodeficiency virus (HIV) infection (HIV antibody positive) 7. Have had or are suffering from other malignant tumors at the same time (except for effectively controlled non melanoma skin basal cell carcinoma, breast/cervical carcinoma in situ, and other malignant tumors that have not been treated and have been effectively controlled in the past five years) 8. Have primary or secondary CNS lymphoma or have a history of CNS lymphoma at the time of recruitment 9. Pregnant and lactating women and childbearing age patients unwilling to take contraceptive measures 10. Those who have a history of drug abuse (use of narcotic drugs or psychotropic drugs for non-medical purposes) or dependence on drugs (sedative hypnotics, analgesics, narcotics, stimulants, and psychotropic drugs, etc.) 11. History of mental illness or cognitive impairment 12. Other investigators judged that it was not suitable to participate in this study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 122 (Estimated)
Dates: Start 2023-04-15 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
relapse rate of T cell lymphoma | three years after transplantation
  relapse rate at three years after transplantation

SECONDARY OUTCOMES:
AEs | from beginning of the conditioning to one month after conditioning
  adverse reactions included gastrointestinal,liver,renal,heart toxicities
immune reconstruction | At 6 months post-transplantation
  the recovery of T, B and NK cells
OS | From date of diagnosis until the end of follow-up or the date of death from any cause, whichever came first，assessed up to 36 months.
  overall survival
PFS | From date of HSCT until the end of follow-up or the date of disease relapse from any cause, whichever came first，assessed up to 36 months.
  progression free survival

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoning Wang, Principal Investigator — First Affiliated Hospital Xi'an Jiaotong University
Locations (1):
- First Affiliated Hospital of Xian Jiaotong University, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: No